CLINICAL TRIAL: NCT00742989
Title: The Short-Term Effect of Osteopathic Lymphatic Treatment on Blood Cell Count, Plasma Protein, and Blood Pressure: A Pilot Study in a Cross-Over Design
Brief Title: Effect of Osteopathic Lymphatic Treatment on Plasma Volume, Protein Concentration and Albumin Concentration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City University of Medicine and Biosciences (Other)
Responsible Party: Patrick G. Clay, PharmD, Director, Dybedal Center for Clinical Research, Kansas City University of Medicine and Biosciences
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: KCUMB-2005-01
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Healthy Volunteers
Keywords: osteopathic; lymphatic; treatment; OLT; normal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): OLT administration
  Interventions: Other: OLT maneuver
- B (Sham Comparator): placebo-OLT
  Interventions: Other: Sham OLT

INTERVENTIONS:
Other: OLT maneuver — direct myofascial release for the thoracic inlet for 30 seconds, supine rib raising for 1 minute on each side of the body, thoracic pumping for one minute, thoracic vacuum for 30 seconds, doming of the abdominal diaphragm for 30 seconds, abdominal pumping for 1 minute, pedal pumping for 1 minute, a second thoracic pump for 1 minute, a second thoracic vacuum for 30 seconds, and a final direct myofascial release for the thoracic inlet lasting 30 seconds
  Arms: A
Other: Sham OLT — Therapeutic massage performed
  Arms: B

SUMMARY:
The goal of this project is to see how much an osteopathic lymphatic treatment (OLT) causes an increase in plasma volume, total plasma protein concentration, and albumin concentration. This is an important step in understanding the effects of OLT, specifically its effects on fluid in the body. The primary role of the lymph system is the return of fluid and proteins lost from the blood vessels. Despite this, no research has been done to see what effects an OLT has on fluid and protein levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy volunteers
* Males
* Age 20 to 40 years

Exclusion Criteria:

* History of cardiovascular, kidney, or liver disease.
* Cannot have taken medication or drugs or have been ill at the time of the study or for two weeks prior.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-05; Primary Completion 2005-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Baseline blood pressure | 15 minute

SECONDARY OUTCOMES:
Plasma proteins | 15 minute

CONTACTS AND LOCATIONS:
Overall Officials: W. Evan Rivers, DO, Principal Investigator — Kansas City University of Medicine and Biosciences; Charlott L. Williiams, RN, CCRC, Study Director — Kansas City University of Medicine and Biosciences; Alan G. Glaros, PhD, Study Director — KCUMB; Kevin Treffer, DO, Study Chair — KCUMB
Locations (1):
- Dybedal Clinical Research Center, Kansas City University of Medicine and Biosciences, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Rivers WE, Treffer KD, Glaros AG, Williams CL. Short-term hematologic and hemodynamic effects of osteopathic lymphatic techniques: a pilot crossover trial. J Am Osteopath Assoc. 2008 Nov;108(11):646-51. PMID 19011227